CLINICAL TRIAL: NCT01639495
Title: THERMOCOOL® SMARTTOUCH™ Catheter for the Treatment of Symptomatic Paroxysmal Atrial Fibrillation Continued Access
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMART-AF CA
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Results first posted 2018-05-15 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-04

CONDITIONS: Drug Refractory Symptomatic Paroxysmal Atrial Fibrillation
Keywords: Drug refractory; Atrial fibrillation; Antiarrhythmic drug failure; Atrial tachyarrhythmias
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This study had a single arm: catheter ablation for PAF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- THERMOCOOL® SMARTTOUCH™ Catheter (Experimental)
  Interventions: Device: THERMOCOOL® SMARTTOUCH™ Catheter

INTERVENTIONS:
Device: THERMOCOOL® SMARTTOUCH™ Catheter — AF Ablation

SUMMARY:
This is a prospective, multicenter, non-randomized continued access clinical evaluation utilizing the THERMOCOOL® SMARTTOUCH™ catheter.

DETAILED DESCRIPTION:
The device is currently under investigation with IDE #G110030. This continued access study will enroll subjects that have participated in the Smart-AF IDE study. Subjects with drug refractory symptomatic paroxysmal atrial fibrillation (PAF) will be considered for this study. Effectiveness and safety endpoints have been defined and will be evaluated post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have had at least 3 atrial fibrillation episodes within 6 months of this study
* Have failed at least one antiarrhythmic drug shown by repeated atrial fibrillation episodes
* 18 years of age or older

Exclusion Criteria including, but not limited to:

* Have had previous ablation for atrial fibrillation
* Have take amiodarone within 6 months of this study
* Have had any heart surgery within the last 60 days
* Have had a heart attack within the last 60 days
* Females who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2014-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Stanford University School of Medicine, Stanford, California
  - Florida Hospital, Orlando, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Loyola University Chicago, Maywood, Illinois
  - University of Kansas Hospitals, Kansas City, Kansas
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - The Valley Hospital, Ridgewood, New Jersey
  - Mt. Sinai School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pennslyvania, Philadelphia, Pennsylvania
  - Texas Cardiac Arrhythmia Foundation, Austin, Texas
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled 148 subjects at 15 clinical sites in the U.S. over the course of approximately 8 months. The first subject was enrolled on July 26, 2012, and the last subject was enrolled on March 18, 2013. The study's last index ablation procedure was on April 24, 2013.
Groups:
- THERMOCOOL® SMARTTOUCH™ Catheter: THERMOCOOL® SMARTTOUCH™ Catheter: Catheter Ablation for Atrial Fibrillation
Period: Overall Study
Arm/Group | THERMOCOOL® SMARTTOUCH™ Catheter
Started | 148 (Patients who signed the informed consent.)
Safety Cohort (Safety population includes those enrolled subjects who underwent insertion of the study catheter.) | 144
Primary Effectiveness Cohort (Safety cohort subjects meeting eligibility criteria & receiving radiofrequency (RF) ablation for AF) | 138
Completed | 132
Not Completed | 16
Not completed — Lost to Follow-up | 6
Not completed — Consented but didn't have study catheter | 4
Not completed — Not meeting inclusion/exclusion criteria | 4
Not completed — No radiofrequency energy applied | 2

BASELINE CHARACTERISTICS:
Population: All subjects who signed informed consent.
Arm/Group | THERMOCOOL® SMARTTOUCH™ Catheter
Number analyzed (Participants) | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All subjects who signed informed consent.
  Participants
    Female | 43
    Male | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All subjects who signed informed consent.
  Participants
    Hispanic or Latino | 2
    Not Hispanic or Latino | 146
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 147
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 148

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieved Freedom From Atrial Tachyarrhythmias
Description: Freedom from documented symptomatic atrial fibrillation/atrial tachycardia/atrial flutter (hereinafter collectively referred to as "atrial tachyarrhythmias") based on electrocardiographic data during the effectiveness evaluation period (Day 91-361). Acute procedure failures, antiarrhythmic drug(AAD) changes and repeat ablation occurring during evaluation period were deemed as primary effectiveness failures
Time Frame: Day 91-361
Population: 137 Study-eligible subjects with per-protocol procedure. CENSORED: 1 lost to follow-up subject without recurrence
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | THERMOCOOL® SMARTTOUCH™ Catheter
Number analyzed (Participants) | 138
Percentage of participants
  Primary Effectiveness Cohort: number analyzed (Participants) | 137
  Primary Effectiveness Cohort | 60.6 [51.9 to 68.8]
  Male: number analyzed (Participants) | 97
  Male | 60.8 [50.4 to 70.6]
  Female: number analyzed (Participants) | 40
  Female | 60 [43.3 to 75.1]
Statistical Analysis 1: Comparison: THERMOCOOL® SMARTTOUCH™ Catheter; Test type: Superiority or Other; Percentage of subjects = 60.6, 95% CI 2-sided [51.9 to 68.8] — The 2-sided 95% confidence intervals are based on exact binomial

2. Secondary Outcome: Peri-procedural Serious Adverse Events
Description: Peri-procedural serious adverse events (SAEs) are those non-primary SAEs occurred within 8-30 days post procedure
Time Frame: Within 8-30 days post procedure
Population: Safety cohort, including Enrolled subjects who underwent insertion of the study catheter.
Measure: Number; unit: Number of participants
Arm/Group | THERMOCOOL® SMARTTOUCH™ Catheter
Number analyzed (Participants) | 144
Number of participants
  Number of subjects had peri-procedural SAEs | 2
  Possibly procedure related | 2
  Not-related to procedure or device | 1

3. Primary Outcome: Incidence of Primary Adverse Events Within Specified Study Period
Description: Primary safety endpoint consists of primary adverse events (AE) within 7 days post procedure Or pulmonary vein stenosis and atrio-esophageal fistula events that occurred within 12 months post-procedure. Primary adverse events include death, myocardial infarction, pulmonary vein stenosis, diaphragmatic paralysis, atrio-esophageal fistula, transient ischemic attack, stroke / cerebrovascular accident, thromboembolism, pericarditis, cardiac tamponade, pericardial effusion, pneumothorax, atrial perforation, vascular access complications, pulmonary edema, initial and prolonged hospitalization (excluding those due to pre-existing arrhythmia recurrence), heart block.
Time Frame: 12 months post procedure
Population: 144 subjects that had study catheter inserted into their body; INCLUDES study ineligible & untreated subjects
Measure: Number (95% Confidence Interval); unit: percentage of subjects with primary AE
Arm/Group | THERMOCOOL® SMARTTOUCH™ Catheter
Number analyzed (Participants) | 144
percentage of subjects with primary AE
  Primary Safety Cohort | 17.4 [11.6 to 24.6]
  Male: number analyzed (Participants) | 102
  Male | 13.7 [7.7 to 22.0]
  Female: number analyzed (Participants) | 42
  Female | 26.2 [13.9 to 42.0]
Statistical Analysis 1: Comparison: THERMOCOOL® SMARTTOUCH™ Catheter; Test type: Superiority or Other; Percentage of subjects with primary AEs = 17.4, 95% CI 2-sided [11.6 to 24.6] — The 2-sided 95% confidence interval is exact binomial

4. Secondary Outcome: Percentage of Subjects Achieved Acute Effectiveness
Description: Acute effectivenesss is defined as confirmation of entrance block into all Pulmonary veins
Time Frame: 5 hours of procedure time
Population: Effectiveness cohort, defined as those enrolled subjects who underwent insertion of the study catheter and an AF ablation procedure. Subjects without RF energy delivery will be excluded (i.e. discontinued subjects).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | THERMOCOOL® SMARTTOUCH™ Catheter
Number analyzed (Participants) | 142
Percentage of participants | 97.2 [95.6 to 98.2]
Statistical Analysis 1: Comparison: THERMOCOOL® SMARTTOUCH™ Catheter; Test type: Superiority or Other; Percentage of subjects = 97.2, 95% CI 2-sided [95.6 to 98.2] — The 2-sided 95% confidence intervals are exact binomial

5. Secondary Outcome: Late Onset Serious Adverse Events
Description: Late onset serious adverse events (SAEs) are those non-primary SAEs occurred after 31 days post procedure
Time Frame: From 31 days post procedure to month 12
Population: Safety cohort, including Enrolled subjects who underwent insertion of the study catheter.
Measure: Number; unit: Number of participants
Arm/Group | THERMOCOOL® SMARTTOUCH™ Catheter
Number analyzed (Participants) | 144
Number of participants
  Number of subjects had late onset SAEs | 27
  Procedure related | 1
  Not-related to procedure or device | 26

ADVERSE EVENTS:
Time Frame: 12 months post procedure
Arm/Group | THERMOCOOL® SMARTTOUCH™ Catheter
Serious Adverse Events (participants affected / at risk) | 46/144
Other Adverse Events (participants affected / at risk) | 40/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THERMOCOOL® SMARTTOUCH™ Catheter (N=144)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 16 (26) — Subjects experienced this serious adervse event required in-patient hospitalization or prolongation of existing hospitalization
Atrial fibrillation (Cardiac disorders) | 4 (4) — Subjects experienced this serious adverse event required in-patient hospitalization or prolongation of existing hospitalization
Atrial flutter (Cardiac disorders) | 3 (3)
Atrioventricular block (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Chest pain (Cardiac disorders) | 2 (2)
Dyspnoea (Cardiac disorders) | 1 (1)
Mitral valve disease (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1)
Pulmonary oedema (Cardiac disorders) | 3 (3)
Abdominal abscess (Gastrointestinal disorders) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 2 (2)
Oesophageal rupture (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Sepsis (Infections and infestations) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 3 (3)
Haematoma (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THERMOCOOL® SMARTTOUCH™ Catheter (N=144)
Fluid overload (Cardiac disorders) | 2 (2)
Oedema peripheral (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Syncope (Cardiac disorders) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Arteriovenous fistula (Vascular disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Chest pain (Cardiac disorders) | 3 (3)
Haematuria (Renal and urinary disorders) | 3 (3)
Pericardial effusion (Cardiac disorders) | 4 (4)
Haematoma (Vascular disorders) | 4 (4)
Arrhythmia (Cardiac disorders) | 19 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator (PI)/Institution and the Sponsor (or its agents) that restricts the PI's rights to discuss, present or publish trial results after the trial is completed. Please contact Biosense Webster, Inc. for additional information.